CLINICAL TRIAL: NCT06268847
Title: Evaluation of the Effect of Marine By-product Hydrolysate Supplementation on the Reduction of Atopic Dermatitis Symptoms : a Randomized, Placebo-controlled, Double-blind Study
Brief Title: Efficacy of Marine By-product Hydrolysate on the Reduction of Atopic Dermatitis Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abyss Ingredients (Industry)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DERMATIDYSS
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: SCORAD; Atopic Dermatitis; Eczema; Hydrolysate; Stress
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo is a capsule with same appearance and organoleptic properties as the active product, containing no active component.
  Interventions: Dietary Supplement: Placebo
- ACT01 (Experimental): The test product is a food supplement presented as a capsule containing a fish hydrolysate.
  Interventions: Dietary Supplement: ACT01
- ACT02 (Experimental): The test product is a food supplement presented as a capsule containing a fish hydrolysate.
  Interventions: Dietary Supplement: ACT02

INTERVENTIONS:
Dietary Supplement: Placebo — The placebo product containing mainly maltodextrin is presented in the same form as the active product, so that people handling the product cannot distinguish between them. The placebo is flavoured in order to have a fishy smell just like the active product.
  2 capsules per day for 90 days of placebo.
  Arms: Placebo
Dietary Supplement: ACT01 — 2 capsules per day (2 per dose) of 300mg (dose per capsule) for 90 days of study product.
  Arms: ACT01
Dietary Supplement: ACT02 — 2 capsules per day (2 per dose) of 300mg (dose per capsule) for 90 days of study product.
  Arms: ACT02

SUMMARY:
This interventional, double-blind, randomized, placebo-controlled study aims to evaluate the effect of a marine by-product hydrolysate supplementation on the reduction of atopic dermatitis symptoms.

DETAILED DESCRIPTION:
The study will be carried out with 108 subjects divided in 3 groups of 36 subjects who will be supplemented with two dosages of the food supplement or a placebo.

This study intends to assess objectively and subjectively the efficacy of a food supplement claimed to improve the skin condition related to atopic dermatitis. The objectives of the study consist in the evaluation of the supplementation to improve the skin condition and symptoms on atopic dermatitis (by SCORAD), to reduce the eczema and severity on atopic dermatitis (by SCORAD and Eczema Area and Severity Index), to reduce the inflammatory signs (by Investigator Global Assessment scale), to moisturize and to improve/maintain the skin barrier.

ELIGIBILITY:
Inclusion Criteria:

* Phototype: I to V;
* Subjects with atopic skin (with at least 1 visible xerosis + inflammation on the body);
* Subjects with a history background of asthma, rhinitis and/or allergic conjunctivitis;
* Subjects with SCORAD between 8 and 30 (at least 50% or more having around 8-10);
* Subjects with BMI between 20 and 30 kg/m2 (limits included);
* Subjects who have not recently participated in another similar study;
* Willingness to take supplements for the duration of the study;
* Willingness not to use products likely to interfere with the test product (collagen, hyaluronic acid, anti-stress products);
* Willingness not to change lifestyle habits;
* Willingness to avoid intensive UV exposure;
* Use of contraception that should not be modified during the study.
* Healthy subject;
* Mentally healthy subject according to Investigator's opinion;
* Subject having given his/her free informed, written consent;
* Subject agrees to taking photograph and then use the image after its pseudonymization;
* Subject willing to adhere to the protocol and study procedures;
* Subject able to understand the study;
* Subject available to attend the study visits.

Exclusion Criteria:

* Pregnant or nursing woman or woman planning to get pregnant during the study;
* Cutaneous marks on the experimental areas, which could interfere with the assessment of skin reactions;
* Subjects who have participated in the last 3 months or are currently participating in another clinical trial that may interfere with the evaluation of the primary endpoint (endpoint AD);
* Current administration of antibiotics;
* Known history of chronic disease such as congenital heart disease, liver or kidney disease, or immune deficiency;
* Topical treatment with immunomodulators (tacrolimus or pimecrolimus) in the three months prior to registration;
* Application of moisturizing products on the experimental area the day of the inclusion of the study;
* Acute or chronic infectious diseases;
* Not meet inclusion criteria;
* Those undergoing aesthetic medicine (fillers, hyaluronic acid injections, botox) that could interference in the experimental area;
* Subjects suffering Alimentary/Eating disorders (i.e. bulimia, psychogenic eating disorders, etc.)
* Subjects having frequent stomach burn;
* Allergy or intolerance to any ingredient of the experimental food supplement;
* Subjects with diabetes mellitus;
* Fish and/or iodine allergy;
* Intestinal conditions or disorders (Crohn's disease, colitis, irritable bowel syndrome, intestinal malabsorption...)
* Recent change, forecast of initiation of an hormonal treatment or change of the usual hormonal treatment during the study or 3 months before the starting of the study;
* Subject having undergone a surgery under general anesthesia within the previous month;
* Exposure in UVA ray sunbed during the 3 months before the start of the study on the experimental area or during the study;
* Subjects protected by the law;
* Subject employed by EUROFINS PRODUCT TESTING, COSMETICS & PERSONAL CARE SPAIN, S.L.U.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
SCORAD (SCORing Atopic Dermatitis) | 12 weeks

SECONDARY OUTCOMES:
EASI (Eczema Area and Severity Index) | 12 weeks
Investigator Global Assessment scale | 12 weeks
  To evaluate the inflammatory signs.
Corneometer | 12 weeks
  To measure skin hydration.
Transepidermal Water Loss (TEWL) | 12 weeks
  To evaluate the epidermal barrier integrity through the transepidermal water loss.
Quality of Life Index - Perceived Stress | 12 weeks
  Auto-questionnaire
Participant's Satisfaction | 12 weeks
  Auto-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DEMILLIERE, MD, Principal Investigator — Dermscan - Eurofins
Locations (1):
- Eurofins, Barcelona, Spain